CLINICAL TRIAL: NCT01423929
Title: Supplemental Oxygen in Catheterized Coronary Emergency Reperfusion
Acronym: SOCCER
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-001452-11
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-02

CONDITIONS: ST Elevation Myocardial Infarction
Keywords: Oxygen; Myocardial infarction; Ambulance; Percutaneous coronary intervention; Cardiac magnetic resonance imaging
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Myocardial Infarction | interventions — Oxygen

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10 L O2/min (Experimental): Oxygen breathing via Oxymask TM
  Interventions: Drug: Oxygen
- Room air (Sham Comparator): Room air breathing via Oxymask TM
  Interventions: Device: Room air

INTERVENTIONS:
Drug: Oxygen — Fitting of Oxymask TM and treatment with 10 L O2/min
  Arms: 10 L O2/min
Device: Room air — Fitting of Oxymask TM
  Arms: Room air

SUMMARY:
The aim of SOCCER is to evaluate the effects of treatment with supplemental O2 before and during acute balloon angioplasty (PCI) for patients with ST-elevation myocardial infarction (STEMI). One hundred STEMI patients are randomized in the ambulance to either standard O2 treatment (10 l/min) or no supplemental O2, to be given until the end of the acute PCI. Cardiac magnetic resonance imaging and echocardiography during the hospital stay is used to assess infarct size and myocardial performance. All patients are followed for 6 months. At 6 months, perceived health and NT-proBNP are recorded for all patients, and an additional echocardiography is performed. The primary endpoint is the fraction of myocardium saved with the acute PCI. The secondary endpoints include the pain difference between inclusion time and start of PCI and myocardial performance on echocardiography.

DETAILED DESCRIPTION:
Almost all patients with ST elevation myocardial infarction (STEMI) in Sweden undergo acute balloon angioplasty (PCI) to open the occluded coronary artery, and thereby to reduce or abolish the myocardial infarction. Standard treatment in these cases is 10-15 l of supplemental oxygen to reduce the myocardial ischemia and the infarct size. It is, however, unknown whether supplemental O2 is beneficial or detrimental to patients with STEMI undergoing PCI.

This study aims to evaluate the effects of treatment with supplemental O2 in acute PCI for STEMI.

The study is a multicenter single blind parallel group randomized trial. One hundred normoxic STEMI ambulance patients accepted for primary PCI are randomized in the ambulance to either standard O2 treatment (10 l/min) or no supplemental O2, to be given until the end of the acute PCI. All patients undergo cardiac MRI at day 4-6 to determine area at risk, infarct size and myocardial salvage index. Fifty patients undergo an extended echocardiography during the hospital stay to assess infarct size and wall motion score index. All patients are followed for 6 months. At 6 months, perceived health (EQ-5D) and NT-proBNP are recorded for all patients, and an additional echocardiography is performed for the subgroup of 50 patients. The primary endpoint is myocardial salvage index. Secondary endpoints include pain difference between inclusion time and start of PCI and wall motion score index on echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* STEMI patient transported with ambulance to SUS Lund or Malmö or Helsingborg hospital, and accepted for acute PCI
* Symptom duration less than 6 hours
* Normal SaO2 (≥ 94 %) measured with pulse oximeter
* Informed consent

Exclusion Criteria:

* Previous AMI
* Inability to make decision to participate; dementia and the like
* For CMR: Significant claustrophobia, prostheses or other magnetic material inside the body

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Myocardial salvage index | Day 4-6 after the acute PCI
  Assessed by cardiac magnetic resonance imaging

SECONDARY OUTCOMES:
Pain difference | At randomization vs at PCI balloon inflation start
  Visual analog scale
Area at risk | Day 4-6 after the acute PCI
  Assessed by cardiac magnetic resonance imaging
Infarct size | Day 4-6 after the acute PCI
  Assessed by cardiac magnetic resonance imaging
Ejection fraction | Day 4-6 after the acute PCI
  Assessed by cardiac magnetic resonance imaging
Microvascular obstruction | Day 4-6 after the acute PCI
  Assessed by cardiac magnetic resonance imaging
Doses of opioids (substance and mg) and betablockers (substance and mg) | Given before and during the PCI
Blood oxygen saturation change | From inclusion to PCI start
  Measured by pulse oximeter
Infarct size | First 24 h after inclusion
  Measured with area under TnT curve
ST segment recovery | 90 minutes after acute PCI
  As measured on ECG
TIMI flow | During acute PCI
  Measured with coronary angiography
Use of heart failure medications (beta blockers, ACEI, ARB, diuretics, digoxin and sinus node inhibitors etc) | At 6 months
Perceived health | At 6 months
  Measured with EQ-5D
Wall motion score index on echocardiography | Day 2-3 after acute PCI
  Measured on echocardiography
Change in wall motion score index | From index hospitalization to 6 months
  Measured on echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Ekelund, MD PhD, Principal Investigator — Skåne University Hospital at Lund
Locations (3):
- Sweden (3):
  - Helsingborg Hospital, Helsingborg
  - SUS Lund, Lund
  - SUS Malmö, Malmo

REFERENCES:
- [Background] Wijesinghe M, Perrin K, Ranchord A, Simmonds M, Weatherall M, Beasley R. Routine use of oxygen in the treatment of myocardial infarction: systematic review. Heart. 2009 Mar;95(3):198-202. doi: 10.1136/hrt.2008.148742. Epub 2008 Aug 15. PMID 18708420
- [Background] Burls A, Cabello JB, Emparanza JI, Bayliss S, Quinn T. Oxygen therapy for acute myocardial infarction: a systematic review and meta-analysis. Emerg Med J. 2011 Nov;28(11):917-23. doi: 10.1136/emj.2010.103564. Epub 2011 Feb 23. PMID 21346260
- [Background] Nicholson C. A systematic review of the effectiveness of oxygen in reducing acute myocardial ischaemia. J Clin Nurs. 2004 Nov;13(8):996-1007. doi: 10.1111/j.1365-2702.2004.00997.x. PMID 15533106
- [Background] Beasley R, Aldington S, Weatherall M, Robinson G, McHaffie D. Oxygen therapy in myocardial infarction: an historical perspective. J R Soc Med. 2007 Mar;100(3):130-3. doi: 10.1177/014107680710000311. No abstract available. PMID 17339308
- [Background] Farquhar H, Weatherall M, Wijesinghe M, Perrin K, Ranchord A, Simmonds M, Beasley R. Systematic review of studies of the effect of hyperoxia on coronary blood flow. Am Heart J. 2009 Sep;158(3):371-7. doi: 10.1016/j.ahj.2009.05.037. Epub 2009 Jul 15. PMID 19699859
- [Derived] Mokhtari A, Akbarzadeh M, Sparv D, Bhiladvala P, Arheden H, Erlinge D, Khoshnood A. Oxygen therapy in patients with ST elevation myocardial infarction based on the culprit vessel: results from the randomized controlled SOCCER trial. BMC Emerg Med. 2020 Feb 18;20(1):12. doi: 10.1186/s12873-020-00309-y. PMID 32070283
- [Derived] Khoshnood A, Akbarzadeh M, Carlsson M, Sparv D, Bhiladvala P, Mokhtari A, Erlinge D, Ekelund U. Effect of oxygen therapy on chest pain in patients with ST elevation myocardial infarction: results from the randomized SOCCER trial. Scand Cardiovasc J. 2018 Apr;52(2):69-73. doi: 10.1080/14017431.2018.1439183. Epub 2018 Feb 13. PMID 29436868